CLINICAL TRIAL: NCT03931395
Title: Evaluation of Honey as Adjunct Therapy to Tylenol and Motrin in Treating Post-Operative Pain and Nausea Following Tonsillectomy
Brief Title: Honey Used as Adjunct Therapy to Tylenol for Post-Op Tonsillectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Katherine Grierson, Registered Nurse, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 190013
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Tonsillectomy
Keywords: Honey; Pediatrics; Post-Operative
MeSH Terms: interventions — Honey; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey Plus Standard of Care (Experimental): The Honey standard of care group will receive treatment as usual, alternating acetaminophen and ibuprofen with a PRN three-day supply of opioid analgesic, plus 1 tsp of honey with every dose of acetaminophen. The Honey standard of care group will receive the first dose of honey in the recovery room with the administration of acetaminophen and will be provided with honey upon discharge.
  Interventions: Dietary Supplement: Honey; Other: Standard of Care
- Standard of Care (Active Comparator): The standard of care group will receive treatment as usual (alternating acetaminophen and ibuprofen with a PRN three-day supply of opioid analgesic).
  Interventions: Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Honey — Will give patients and families included in the honey standard of care group 40 packets of hospital approved honey to implement in the tonsillectomy post-operative care of the child
  Arms: Honey Plus Standard of Care
Other: Standard of Care — Patients will receive standard post operative medications per surgeon

SUMMARY:
Tonsillectomies are the second most common surgery with over half a million procedures in the United States for 2006. Tonsillectomies are considered a painful surgical procedure performed on children resulting in pain and nausea/vomiting for up to 7 days postoperatively. Up until recently, doctors have been prescribing upwards of ten days' worth of opioid pain medication for children following tonsillectomies due to the high incidence of pain expected afterwards. Effective July 1st, 2018, new laws regarding opioid restrictions came into place that restricted doctor's abilities to write for more than three days' worth of opioid pain medication without having to fill out sizeable amounts of additional paperwork. This law was put in place to combat the ongoing opioid epidemic that plagues this country. What the investigators are left with for the treatment of pain following these procedures are simply Tylenol and Motrin with a limited amount of opioid. With this being considered a highly painful surgery with a difficult recovery, more options are needed to effectively treat pain and reduce the incidence of emergency room visits and phone calls to the clinic regarding pain control in the postoperative period.

Studies in Europe have shown that honey is an effective adjunct treatment option in the reduction of pain in pediatric postoperative tonsillectomies. These studies are few and far between and more research needs to be conducted to validate these claims particularly in the United States where research on this subject has been extremely limited. Further, the extent to which families and health care providers in the United States would be receptive to using honey for children's postoperative pain is unclear since honey is considered a complementary and alternative medicine (CAM) intervention.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking families
* male or female
* 2-17 years old undergoing a routine tonsillectomy procedure.
* English speaking families in the waiting room whose children are having any type of surgery during the time period we are enrolling the tonsillectomy patients.

Exclusion Criteria:

* Subjects will be excluded for any of the following reasons: Any child undergoing or has already undergone a tonsillectomy who has a genetic syndrome or developmental disability (e.g., Trisomy 21, Angelman Syndrome, etc.) which could impact the course of postoperative pain management.
* Any child who has an allergy to honey.
* Non English speaking families.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Pain scores as assessed by the Numerical Rating scale in participants who are given honey. | Baseline to 3 weeks
  Parents will use the Numerical Rating scale to assess their Childs pain. The range is 0-10, 0=No pain and 10 = Worst pain ever. This scale is used for patients who are developmentally able (ages 9 and up)
Pain scores as assessed by the Wong-Baker FACES scale in participants who are given honey. | Baseline to 3 weeks
  Parents will use the FACES pain scale. They will have the child choose between a range of faces that indicate a pain score of 0-10, 0 (a smiling face) = no pain and 10 (crying face) = worst pain ever. This scale is used for patients who are developmentally able (ages 3-9)
Pain scores as assessed by the FLACC scale in participants who are given honey. | Baseline to 3 weeks
  Parents will use use the FLACC pain scale, 0 = No pain and 10 = Worst pain ever. This scale will be used in children who developmentally can not rate their own pain (ages 2 months to 7 years)
Pain scores as assessed by the Numerical Rating scale in participants who receive standard of care (Tylenol, motoring & oxycodone). | Baseline to 3 weeks
  Parents will use the numerical rating scale to assess their Childs pain. The range is 0-10, 0=No pain and 10 = Worst pain ever. This scale is used for patients who are developmentally able (ages 9 and up)
Pain scores as assessed by the Wong-Baker FACES scale in participants who receive standard of care (Tylenol, motoring & oxycodone). | Baseline to 3 weeks
  Parents will use the FACES pain scale. They will have the child choose between a range of faces that indicate a pain score of 0-10, 0 (a smiling face) = no pain and 10 (crying face) = worst pain ever. This scale is used for patients who are developmentally able (ages 3-9)
Pain scores as assessed by the FLACC scale in participants who receive standard of care (Tylenol, motoring & oxycodone). | Baseline to 3 weeks
  Parents will use use the FLACC pain scale, 0 = No pain and 10 = Worst pain ever. This scale will be used in children who developmentally can not rate their own pain (ages 2 months to 7 years)
Nausea scores as assessed by the baxter barf scale in participants who receive honey. | Baseline to 3 weeks
  Parents will use the baxter barf scale by selecting or having their child select a face that represents nausea on a scale of 0 to 10, 0 = no nausea and 10 = actively vomiting.
Nausea scores as assessed by the baxter barf scale in participants who receive standard of care. | Baseline to 3 weeks
  Parents will use the baxter barf scale by selecting or having their child select a face that represents nausea on a scale of 0 to 10, 0 = no nausea and 10 = actively vomiting.

SECONDARY OUTCOMES:
Beliefs and receptiveness of patient families to complementary and alternative medicine (CAM) and use of honey. | Baseline to 3 weeks
  Families will be given a CAM questionnaire to complete. The questionnaire asks families to rate on a scale of strongly disagree to strongly agree and asks questions like "The more knowledge a person has about CAM, the more likely they are to use it" and "There are less side effects when taking natural remedies" Families who select strongly disagree = they definitely do not agree with the statement. If they select strongly agree = they very much agree with the statement. Families will get this survey at the beginning of the study and get it again at the end to evaluate if their statement responses have changed.
  The beliefs and attitudes toward CAM were measured based on a 7-point Likert scale, with 1 representing strongly agree and 7 representing strongly disagree; mean scores and standard deviation were calculated for each of the 13 items.
The relation between the beliefs and receptiveness of nursing staff to complementary and alternative medicine (CAM) and use of honey. | Baseline to 3 weeks
  Nursing staff will receive a voluntary survey containing the CAM belief scale. The survey asks nurses to rate on a scale of Strongly disagree to Strongly agree and asks questions such as "I assess my patient for CAM use" or "I believe that CAM has a role in my practice." Strongly disagree = they definitely do not agree with the statement, strongly agree = They strongly agree with the statement.
  The beliefs and attitudes toward CAM were measured based on a 7-point Likert scale, with 1 representing strongly agree and 7 representing strongly disagree; mean scores and standard deviation were calculated for each of the 13 items.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Card, MSN, Study Director — Nursing Research Consultant
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaryszak EM, Lander L, Patel AK, Choi SS, Shah RK. Prolonged recovery after out-patient pediatric adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2011 Apr;75(4):585-8. doi: 10.1016/j.ijporl.2011.01.024. Epub 2011 Feb 15. PMID 21324535
- [Background] Ozlugedik S, Genc S, Unal A, Elhan AH, Tezer M, Titiz A. Can postoperative pains following tonsillectomy be relieved by honey? A prospective, randomized, placebo controlled preliminary study. Int J Pediatr Otorhinolaryngol. 2006 Nov;70(11):1929-34. doi: 10.1016/j.ijporl.2006.07.001. Epub 2006 Aug 17. PMID 16914210
- [Background] Boroumand P, Zamani MM, Saeedi M, Rouhbakhshfar O, Hosseini Motlagh SR, Aarabi Moghaddam F. Post tonsillectomy pain: can honey reduce the analgesic requirements? Anesth Pain Med. 2013 Summer;3(1):198-202. doi: 10.5812/aapm.9246. Epub 2013 Jul 1. PMID 24223362
- [Background] Bardy J, Slevin NJ, Mais KL, Molassiotis A. A systematic review of honey uses and its potential value within oncology care. J Clin Nurs. 2008 Oct;17(19):2604-23. doi: 10.1111/j.1365-2702.2008.02304.x. PMID 18808626
- [Background] Abdullah B, Lazim NM, Salim R. The effectiveness of Tualang honey in reducing post-tonsillectomy pain. Kulak Burun Bogaz Ihtis Derg. 2015;25(3):137-43. doi: 10.5606/kbbihtisas.2015.00008. PMID 26050853
- [Background] Mohebbi S, Nia FH, Kelantari F, Nejad SE, Hamedi Y, Abd R. Efficacy of honey in reduction of post tonsillectomy pain, randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2014 Nov;78(11):1886-9. doi: 10.1016/j.ijporl.2014.08.018. Epub 2014 Aug 21. PMID 25193590
- [Background] Gedaly-Duff V, Ziebarth D. Mothers' management of adenoid-tonsillectomy pain in 4- to 8-year-olds: a preliminary study. Pain. 1994 Jun;57(3):293-299. doi: 10.1016/0304-3959(94)90004-3. PMID 7524009
- [Background] Finley AG, McGrath PJ, Forward PS, McNeill G, Fitzgerald P. Parents' management of children's pain following 'minor' surgery. Pain. 1996 Jan;64(1):83-87. doi: 10.1016/0304-3959(95)00091-7. PMID 8867249
- [Background] Gabalski EC, Mattucci KF, Setzen M, Moleski P. Ambulatory tonsillectomy and adenoidectomy. Laryngoscope. 1996 Jan;106(1 Pt 1):77-80. doi: 10.1097/00005537-199601000-00015. PMID 8544633